CLINICAL TRIAL: NCT02634229
Title: Constitution of a Cohort of Families With Monogenic Diabetes to Identify Novel Causes of Non Auto-immune Diabetes Mellitus in Children and Young Adults
Brief Title: Predisposition Genes in Monogenic Diabetes (DIAMONO)
Acronym: DIAMONO
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: NI11010
Record Dates: First submitted 2015-10-05; First posted 2015-12-17 (Estimated); Last update posted 2016-02-17 (Estimated); Status verified 2015-08

CONDITIONS: Non Autoimmune Monogenic Diabetes
Keywords: monogenic diabetes; MODY; beta-cell; insulin secretion
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Diabetic family members: (i) probands negative for GCK/MODY2 , HNF1A/MODY3 genes and HNF4A/MODY1; (ii) dominant inheritance of diabetes (three consecutive affected generations, or two generations with at least 2 diabetic patients in a generation); (iii) Diagnosis of diabetes before age 40 years in at least 3 diabetic family members; (iv) negative testing for anti-GAD and IA2-antibodies; and (v) body mass index < 30 kg/m2 (to avoid inclusion of patients with insulin-resistant type 2 diabetes).
  Interventions: Genetic: blood sample
- Healthy relatives: Healthy subjects whose relationship is relevant for genetic analysis and necessary for the validation step (family cosegregation study)
  Interventions: Genetic: blood sample

INTERVENTIONS:
Genetic: blood sample

SUMMARY:
Monogenic diabetes accounts for 1-2% of diabetes cases, although it is often misdiagnosed as either type 1 diabetes or type 2 diabetes. Knowledge of the genetic etiology of diabetes enables more appropriate treatment, better prediction of disease progression, screening of family members and genetic counseling. These monogenic diabetes result from gene mutations that reduce beta-cell function. To date, about 20 genes involved in insulin-secretion pathway hav been identified; they correspond to a broad of two main clinical conditions [neonatal diabetes mellitus (NDM) and Maturity-Onset Diabetes of the Young (MODY)]. However, it still remains subtypes of monogenic diabetes that are unelucidated. The investigators project focus on families with a clinical and familial history highly suggesting a MODY diabetes but without genetic etiology. The investigators objective is to set up a collection of families with at least three family members presenting a MODY diabetes.

DETAILED DESCRIPTION:
There are several monogenic disorders of pancreatic beta-cell function, characterized by various degrees of chronic hyperglycemia. They are usually diagnosed early in life, in neonates or during infancy, childhood or even in young adults. These diseases comprise a broad spectrum of diabetic phenotypes including neonatal diabetes mellitus (NDM), non auto-immune diabetes in infancy, dominantly inherited forms of early-onset diabetes [also named Maturity-Onset Diabetes of the Young (MODY)] and very rare diabetes-associated syndromes.

So far, causal mutations in more than 20 genes that are highly expressed in the pancreatic beta-cells have been identified in NDM and MODY. These discoveries have demonstrated several aetiological mechanisms of beta-cell dysfunction that are involved in distinct subtypes of monogenic diabetes, including reduced beta-cell number or development (as for mutations in PDX1, PTF1A, HNF1B), reduced glucose sensing and metabolism (mutations in GCK, INS, HNF1A, HNF4A), failure of membrane depolarization (mutations in KCNJ11, ABCC8) and increased destruction of the beta-cell (mutations in INS, EIF2AK3, WFS1), which result in inadequate insulin secretion despite a chronic hyperglycemia. Additional unknown MODY loci may be responsible for 20-30% of the early-onset diabetes cases with a dominant pattern of inheritance, and a proportion of 50% of the NDM/MDI patients are still unelucidated, suggesting that defects in further pathways in the insulin-secreting beta-cell are responsible for monogenic diabetes.

The investigators project is to collect of 15 MODY-X families. This collection will allow the search of novel genes involved in MODY diabetes. The establishment of the cohort will be based on the recruitment of families of MODY-X probands analyzed in the Department of Genetics (Pitie-Salpetriere hospital). This laboratory performs the genetic testing of MODY. To select families eligible to that project, the investigators will apply the following criteria : (i) probands negative for GCK/MODY2 , HNF1A/MODY3 genes and HNF4A/MODY1; (ii) dominant inheritance of diabetes (three consecutive affected generations, or two generations with at least 2 diabetic patients in a generation); (iii) Diagnosis of diabetes before age 40 years in at least 3 diabetic family members; (iv) negative testing for anti-GAD and IA2-antibodies; and (v) body mass index < 30 kg/m2 (to avoid inclusion of patients with insulin-resistant type 2 diabetes).

The investigators will collect clinical information for the selected cases and families of interest according to a standardized questionnaire.

DNA samples will be collected for diabetic family members and healthy relatives. All will sign an informed written consent.

ELIGIBILITY:
Inclusion Criteria:

* No mutations in known genes associated with MODY (GCK, HNF1A, HNF4A)
* ≥ 3 cases of diabetes in the family over several generations
* An age at diagnosis of diabetes <40 years for 3 subjects diabetics in the family
* Absence of anti-GAD and anti-A2 of antibodies
* No argument for type 2 diabetes

Exclusion Criteria:

* Diabetic subjects
* Healthy subjects whose relationship is relevant for genetic analysis and necessary for the validation step (family cosegregation study)
* These subjects will be over the age of 18, affiliated to a social protection scheme or copyright holder and will signed an informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Diabetic family members and healthy relatives
Sampling Method: Non-Probability Sample
Enrollment: 96 (Actual)
Dates: Start 2012-09; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Identification of novel predisposition gene | 1 day
  Identification of pathogenic mutations segregating with the "diabetes" phenotype and absent in unaffected relatives.

SECONDARY OUTCOMES:
Correlation between genotype and age at diagnosis | 1 day
Correlation between genotype and BMI | 1 day
Correlation between genotype and treatment | 1 day
Correlation between genotype and mode of presentation | 1 day
Correlation between genotype and complications of diabetes | 1 day
Correlation between genotype and fasting plasma glucose | 1 day
Correlation between genotype and HbA1c | 1 day
  at diagnosis and at last examination

CONTACTS AND LOCATIONS:
Overall Officials: Christine BELLANNE-CHANTELOT, PharmD-PhD, Study Director — Assistance Publique - Hôpitaux de Paris